CLINICAL TRIAL: NCT01215656
Title: Effect of a Follow on Formula With Lactobacillus Fermentum on the Incidence of Infections
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Puleva Biotech (Industry)
Responsible Party: Federico Lara Villoslada, Puleva Biotech
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: L. fermentum infections
Record Dates: First submitted 2010-10-05; First posted 2010-10-06 (Estimated); Last update posted 2010-10-07 (Estimated); Status verified 2010-10

CONDITIONS: Incidence of Infectious Diseases
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Probiotic (Experimental): follow on formula with the probiotic Lactobacillus fermentum
  Interventions: Dietary Supplement: Lactobacillus fermentum
- Control (Active Comparator): follow on formula without probiotics
  Interventions: Dietary Supplement: Follow on formula without probiotics

INTERVENTIONS:
Dietary Supplement: Lactobacillus fermentum
  Arms: Probiotic
Dietary Supplement: Follow on formula without probiotics
  Arms: Control

SUMMARY:
The objective of the study is to evaluate the effects of a follow on formula containing the human milk probiotic Lactobacillus fermentum on the incidence of infection in 6 months old infants.

ELIGIBILITY:
Inclusion Criteria:

* 6 months old children born at term
* written consent from parents

Exclusion Criteria:

* frequent gastrointestinal disorders (frequent diarrhoeas, constipation episodes, gastroesophageal reflux)
* gastrointestinal surgery
* cow's milk protein allergy
* metabolic diseases (diabetes or lactose intolerance)
* immune deficiency
* antibiotic treatment during the trial and/or recent (within the preceding 3 weeks)

Ages: 6 Months to 7 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 188 (Actual)
Dates: Start 2008-05; Primary Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Incidence of infectious diseases

REFERENCES:
- [Derived] Maldonado J, Canabate F, Sempere L, Vela F, Sanchez AR, Narbona E, Lopez-Huertas E, Geerlings A, Valero AD, Olivares M, Lara-Villoslada F. Human milk probiotic Lactobacillus fermentum CECT5716 reduces the incidence of gastrointestinal and upper respiratory tract infections in infants. J Pediatr Gastroenterol Nutr. 2012 Jan;54(1):55-61. doi: 10.1097/MPG.0b013e3182333f18. PMID 21873895